CLINICAL TRIAL: NCT03364569
Title: Usefullness of Peri-operative Tranexamic Acid in Primary Breast Augmentation With Implants.
Acronym: DRAINAGE
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD2315
Record Dates: First submitted 2017-11-24; First posted 2017-12-06 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Plastic Surgery
Keywords: Drainage; Breast augmentation; Tranexamic acid
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participant with tranexamic acid.: The investigators followed the recommendations of one gram, two times a day, starting at the end of the surgery so as to avoid any adverse effects. The participants received two grams of Spotof ® (C.C.D laboratory, Portugal) as an oral liquid solution during three days.
  Interventions: Procedure: Tranexamic acid
- Participant without tranexamic acid.: This group concerns participants followed without acid tranexamic treatment. Investigators will observe the postoperative practices and complications observed, according to the surgical habits.

INTERVENTIONS:
Procedure: Tranexamic acid — Participants with taking tranexamic acid (2 x 1g per day) as a preventive and without adjuvant treatment.
  Groups: Participant with tranexamic acid.

SUMMARY:
Tranexamic acid (TXA), as an antifibrinolytic agent, has shown a tremendous interest in surgery by reducing blood loss ; but only few articles have been reported in the plastic surgery scope. The aim of this study was to investigate whether oral administration of TXA reduces surgical drainage in primary breast augmentation using implants.

DETAILED DESCRIPTION:
A total of forty participants were included in this case-control study over a fifteen months period. The participants were divided in two equal groups. The case group (TXA group) was treated with a daily oral administration of two grams of tranexamic acid whereas the control group (noTXA group) was not treated. The data that has been recorded is the gender, the age, the implant volume (cc), the shape of the implant (round or anatomical), the type of surgical pocket (pre-muscular or retro-muscular), the texture of the implant (textured or smooth), the operating time (in minutes), the blood pressure operative average during surgery, volume of fluid daily (right and left) and complications (hematoma, infection, deep vein thrombosis, pulmonary embolism, anaphylaxis and early exposure to implants).

Three investigators were enrolled in the study, including the corresponding author. Two investigators performed the intervention, operating one breast each.

At the end of the surgical procedure, a drain was put in the retro-pectoral space on each breast side. A compressive garment was immediately fitted before the exit of the participant. The participants received oral analgesics according to the hospital guidelines and no thromboprophylaxis was given, as it is a standard recommendation of the French Society of Anaesthesiologists (SFAR).

Oral administration of the TXA had never been tested in breast augmentation indications, and the investigators followed the recommendations of one gram, two times a day, starting at the end of the surgery so as to avoid any adverse effects. The participants received two grams of Spotof ® (C.C.D laboratory, Portugal) as an oral liquid solution during three days.

All participants were interviewed by a nurse every four hours starting at the end of the post-operative recovery room till the exit of their hospital stay. Drain fluid volume in the vacuum devices was recorded every twenty four hours. The drains were removed when production was below forty milliliter per twenty four hours, according to hospital routine. Any early (less than seven days) or late (better than thirty days) post-operative complications were also listed. All participants had a consultation seven days and two months after the surgery according to the department guidelines. A hotline telephone number has been given to participants to facilitate contact if any inconvenient consequences have occurred.

In each sub-group (no TXA and TXA), the main outcome was the drain fluid production during the study which was registered for each breast every twenty four hours after the surgery and at the exit of the participant. Volume were stored and collected in milli-liters (mL) without consistency or color analysis. The age (in years), the implant volume (in milliliters), the shape (round or anatomic) and the texture (smooth or textured), the mean operative time (in minutes), the mean operative arterial pressure (in mmHg) were also recorded as well as the length of the hospital stay (in days). Any surgical complications and any side effects associated to the TXA drug were also listed.

ELIGIBILITY:
Inclusion Criteria:

* Woman with Primary Breast Augmentation

Exclusion Criteria:

* Past History of Thromboembolism
* Use of anticoagulant or platelet-inhibiting drugs
* Severe Co-morbidity (ASA III)
* Pre-pectoral Implant Pocket Location
* Breast lipofecting

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Breast augmentation with placement of prosthetic implants.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Post-operative drainage volume | Through study completion, an average of 2 years.
  At the end of the surgical procedure, a drain was put in the retro-pectoral space on each breast side. A compressive garment was immediately fitted before the exit of the patient. The participants received oral analgesics according to the hospital guidelines and no thromboprophylaxis was given, as it is a standard recommendation of the French Society of Anaesthesiologists (SFAR). Drain fluid volume in the vacuum devices was recorded every 24 hours. The drains were removed when production was below 40 mL per 24h, according to hospital routine. Volume were stored and collected in milli-liters (mL) without consistency or color analysis. Age (in Years), Implant Volume (in milli-liters), Shape (Round or Anatomic) and Texture (Smooth or Textured), Mean Operative Time (in minutes), Mean Operative Arterial Pressure (in mmHg) were also recorded as well as the length of the Hospital Stay (in Days).

SECONDARY OUTCOMES:
Post-operative complications | Through study completion, an average of 2 years.
  The investigators observed postoperative complications. All participant were interviewed by a nurse every 4 hours starting at the end of the post-operative recovery room till the exit of their hospital stay. Any early (< 7 days) or late (> 30 days) post-operative complications were also listed. All the participants had a consultation 7 days and 2 months after the surgery according to the department guidelines. A Hotline phone number was given to the patients to ease contact if any inconvenient aftermath occured. Any surgical complications and any side effects associated to the TXA drug were also listed.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas COLSON, Principal Investigator — Hôpital NOVO

IPD SHARING:
Plan to Share IPD: No